CLINICAL TRIAL: NCT04020497
Title: Ensemble Programme an Early Intervention for Informal Caregivers of Psychiatric Patients: a Randomized Controlled Trial
Brief Title: Ensemble Programme an Early Intervention for Informal Caregivers of Psychiatric Patients
Acronym: Ensemble
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institut et Haute Ecole de la Santé la Source (Other)
Responsible Party: Principal Investigator, Shyhrete Rexhaj, Porfessor associate HES, Institut et Haute Ecole de la Santé la Source
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EnsembleRCT
Record Dates: First submitted 2019-07-12; First posted 2019-07-16 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Psychological Distress
Keywords: target support; informal caregiver; recovery; well-being; burden; quality of life
MeSH Terms: interventions — Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ensemble + SAU (Support as usual) (Experimental): The five-session Ensemble program provided to informal caregivers targeted support + SAU
  Interventions: Behavioral: Ensemble programme; Other: SAU
- SAU (Support as usual) (Active Comparator): SAU alone which was chosen as a control condition.
  Interventions: Other: SAU

INTERVENTIONS:
Behavioral: Ensemble programme — Ensemble is a individualized programme to address informal caregiver's specific unmet needs, emotions and social resources, in order to offer a targeted support in five sessions.
  Other Names: Ensemble
  Arms: Ensemble + SAU (Support as usual)
Other: SAU — Informal caregivers have often to manage the situation in usual different ways. Support as usual (SAU) alone consists of an informal support by patient's clinical team. Specific psychoeducational programs depending on patient's illnes (like "Profamille" for schizophrenia) or peer-support depending to the voluntary work of families' associations. Some general professional services focused on informal caregivers or relatives in order to inform and orient them if they are avaible in the study area. No attempts have been made to standardize this treatement as SAU depend to informal caregiver's need and knowledge of the health system, also her/his capacity or possibility to be in contact with patient's clinical team.
  Other Names: Support as usual

SUMMARY:
This study focuses on the difficulties of maintaining optimal psychological health and quality of life for caregivers in adult psychiatry while they play an important role in helping patients with severe psychiatric disorders. It evaluates the addition of a 5 session psychological program, named Ensemble. Half of the participants will receive their usual support and Ensemble in combination, while the other half will receive usual support only.

DETAILED DESCRIPTION:
The recent statistics showed that mental disorders affect one in four people in the world. In this context, informal caregivers are key actors in the health care system through their support. This support can be associated with very high burden and distress. Informal caregivers can experience serious situations with potential negative consequences on their quality of life, their own health and the health of patients. Data recommended to intervene at the onset of disease to improve the impact of an intervention. It seems important also to intervene while the patient is in an acute phase of illness to better support informal caregivers' emotional needs. In addition, providing emotional support for informal caregivers at the beginning of an illness in particular is recommended because this is a critical phase. The experience of painful emotions, such as denial of disease and feelings of being overwhelmed or shocked can have serious consequences on their health and on the patient's recovery. Previous studies identified that informal caregivers need tailored knowledge about the patient's illness, clarification about their roles and responsibilities, better control over their own life and effective collaboration with health professionals. Most of the interventions published in the literature focus on the ill family member and its support but not on the specific needs of the informal caregivers as the core intervention. To reduce the gap between scientific recommendations and actual practice, the investigators developed, tailored and tested a new intervention called Ensemble.

Ensemble is a brief individualized intervention designed to promote the well-being of informal caregivers who experience the effects of patients' psychiatric disorders. The five-session Ensemble program provided to informal caregivers targeted support to address their specific unmet needs, emotions and social resources. A professional addressed this programme to the informal caregiver delivered independently of the patient's treatment.

Ensemble assesses the needs of informal caregivers and provides a tailored brief support. Results of a pilot study showed that psychological health and optimism of informal caregivers were improved. For these reasons, there is a clear research and clinical need to establish whether Ensemble programme is clinically effective by using a randomized, controlled, and assessor-blind trial. A combination of Ensemble plus support as usual (SAU) will be compared to SAU alone. Informal caregivers of individuals suffering from mental disorders will undergo either intervention for five sessions, during a six weeks average time. Measure will assess participants' current psychological health state and optimism. These different measures will be performed at the time of inclusion, at the end of the intervention, and at two months follow-up. At the end of the program, individual qualitative structured interviews will be performed to assess acceptability of the programme.

ELIGIBILITY:
Inclusion Criteria:

* Being at least 18 years old
* Living in the French-speaking cantons of Switzerland (commonly referred to as "Romandy")
* Speaking French
* Having an adult relative suffering from a psychiatric disorder (with or without an established diagnosis)
* Having the capacity to agree to participate in the project

Exclusion Criteria:

- Having les than 20 on the Zarit score.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Psychological state change on the Global Severity Index (GSI) | Change from Baseline composite on the GSI score at post-test, and at 2 months follow
  Assessment of psychological symptoms and psychological distress (BSI scale). The Brief Symptom Inventory (BSI) includes 53 items organized into 9 primary and clinically relevant symptom dimensions: 1) somatization, 2) obsessive-compulsive, 3) interpersonal sensitivity, 4) depression, 5) anxiety, 6) hostility, 7) phobic anxiety, 8) paranoid ideation and 9) psychoticism. This scale has also three global distress indices: The Global Severity Index (GSI), the Positive Symptom Distress Index (PSDI) and the Positive Symptom Total (PST).

SECONDARY OUTCOMES:
Optimism change on the Life Orientation Test-Revised (LOT-R) | Change from Baseline total score of the LOT-R at post-test, and at 2 months follow
  Assessement of optimism level (LOT-R scale). The Life Orientation Test - Revised (LOT-R) measures an individual's optimism regarding a given situation. This scale measure the adaptive strategies correlated with well-being. This scale includes 10 items; three items measure optimism, three other measure pessimism, and four of the 10 items function as fillers.
Quality of life change on the Mental Component Score (MCS) | Change from Baseline composite on the MCS score at post-test, and at 2 months follow
  Assessment of the quality of life (36-item Medical Outcome Study Short-Form Health Survey (SF-36)). This scales measures some health indicators related to the quality of life. It includes 36 items and permitted, in clinical and general population settings, to evaluated eight health dimensions: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. Two global scores, i) A Physical Component Score (PCS) and ii) the Mental Component Score (MCS) obtained by grouping the eight dimensions permit to have global variables.
Burden level change on the Zarit Burden Intervieuw (ZBI) | Change from Baseline on the Zarit score at post-test and at 2 months follow
  Assessment of the informal caregiver's burden level by the Zarit Burden Interview. This 22-item scale assesses the subjective burden (emotional, physical and financial) for an informal caregiver of an individual with loss of autonomy.
Standardized severity of the patient's illness change on the Social an Occupational Functioning Assessment Scale (SOFAS) | Change from Baseline on the SOFAS score at 2 months follow
  Assessment of the severity patient's illness mesured by Social and Occupational Functioning Assessment Scale (SOFAS) and completed by the informal caregiver. The SOFAS is a scale from 0 to 100 demonstrating the patient's social functioning. In this study, this score will be measured according to the informal caregiver's representation.

CONTACTS AND LOCATIONS:
Overall Officials: Shyhrete Rexhaj, Principal Investigator — Institut et Haute école de la Santé, La Source
Locations (1):
- La Source, School of Nursing Sciences, HES-SO University of Applied Sciences Western Switzerland, Lausanne., Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rexhaj S, Leclerc C, Bonsack C, Favrod J. Approche pour cibler le soutien auprès des proches aidants de personnes souffrant de troubles psychiatriques sévères. Annales Médico-psychologiques, revue psychiatrique 75 (9): 781-788. 2017.
- [Background] Rexhaj S, Monteiro S, Golay P, Coloni-Terrapon C, Wenger D, Favrod J. Ensemble programme for early intervention in informal caregivers of psychiatric adult patients: a protocol for a randomised controlled trial. BMJ Open. 2020 Jul 30;10(7):e038781. doi: 10.1136/bmjopen-2020-038781. PMID 32737097
- [Result] Rexhaj S, Leclerc C, Bonsack C, Golay P, Favrod J. Feasibility and Accessibility of a Tailored Intervention for Informal Caregivers of People with Severe Psychiatric Disorders: a Pilot Study. Front Psychiatry. 2017 Sep 21;8:178. doi: 10.3389/fpsyt.2017.00178. eCollection 2017. PMID 28983262
- [Derived] Rexhaj S, Martinez D, Golay P, Coloni-Terrapon C, Monteiro S, Buisson L, Drainville AL, Bonsack C, Ismailaj A, Nguyen A, Favrod J. A randomized controlled trial of a targeted support program for informal caregivers in adult psychiatry. Front Psychiatry. 2023 Nov 30;14:1284096. doi: 10.3389/fpsyt.2023.1284096. eCollection 2023. PMID 38098635